CLINICAL TRIAL: NCT01424969
Title: Effects of Platelet-Rich Fibrin Matrix on Repair Integrity of At-Risk Rotator Cuff Tears
Brief Title: The Effects of Platelet Rich Plasma on the Integrity of Rotator Cuff Repair
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Robert Burks, MD, University of Utah
Other Study IDs: 29598
Record Dates: First submitted 2011-08-22; First posted 2011-08-29 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Rotator Cuff Tear Arthropathy
Keywords: rotator cuff repair; arthroscopic; platelet-rich plasma; platelet-rich fibrin matrix; outcomes; tendon healing; magnetic resonance imaging
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PRFM Group: Patients were selected prospectively for the study based on a 3-part algorithm used to identify rotator cuff tears at risk for retear. A total algorithm score of 3 or greater was required for enrollment in the study.
- Control Group: The control group were recruited retrospectively. Patients who have undergone arthroscopic repair of rotator cuff tears with similar size characteristics without PRFM augmentation will be encouraged to participate by letter initially, and then by telephone invitation. The same inclusion and exclusion criteria applied. MRI, pain, and functional scores will be collected in the same manner as the PRFM group at one time point at least one year post operatively.

SUMMARY:
The purpose of this study was to determine the effect of platelet-rich fibrin matrix (PRFM) augmentation to at-risk arthroscopic rotator cuff repairs on healing rates and functional outcome scores. The investigators performed an observational cohort study in which a consecutive series of patients with rotator cuff tears at risk for retear was prospectively evaluated after arthroscopic repair augmented with PRFM. Clinical and magnetic resonance imaging (MRI) outcomes of the PRFM-augmented repairs were compared with historical controls with similar at-risk tears without PRFM augmentation.

DETAILED DESCRIPTION:
Increased age, larger tear size, and more advanced fatty degeneration of the rotator cuff musculature have been correlated with poorer healing rates after rotator cuff repair. Platelets are an endogenous source of growth factors present during rotator cuff healing.

The investigators hypothesis is that augmentation of rotator cuff repairs with platelet-rich fibrin matrix (PRFM) may improve the biology of rotator cuff healing and thus improve functional outcome scores and retear rates after repair.

Rotator cuff tears at risk for retear were prospectively identified using an algorithm; points were assigned for age (50-59 years = 1; 60-69 years = 2; .70 years = 3), anterior-to-posterior tear size (2-2.9 cm = 0; 3-3.9 cm = 1; .4 cm = 2), and fatty atrophy (Goutallier score 0-2 = 0; Goutallier score 3-4 = 1). Three points were required for enrollment. Arthroscopic rotator cuff repair was performed with the addition of PRFM. Preoperative and 1-year postoperative magnetic resonance imaging (MRI) and functional outcome scores were obtained. Imaging and functional outcomes were compared with historical controls meeting the same enrollment criteria.

Enrollment for the study began in September 2008 and continued until March 2010.

ELIGIBILITY:
Inclusion Criteria:

* Algorithm score greater and equal to 3
* Both men and women over the age of 50
* Full-thickness rotator cuff tear at least 2 cm in size
* Tear repairable by arthoscopic-only techniques

Exclusion Criteria:

* Inflamation joint disease
* Active use of oral steroids
* Irreparable rotator cuff tear
* Subscapularis tear requiring open repair
* Claustrophobia
* Prior rotator cuff sugery on the affected shoulder
* Failure to return for follow-up magnetic resonance imaging scan

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic rotator cuff tears identified by clinical exam and MRI that measure greater than two centimeters or are retracted medially to the level of the humeral head cartilage that meet the inclusion/exclusion criteria were asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Preoperative and 1-year postoperative magnetic resonance imaging (MRI) and functional outcome scores | 1 year
  Patients with symptomatic rotator cuff tears identified by clinical exam and MRI that measure greater than two centimeters or are retracted medially to the level of the humeral head cartilage. Shoulder pain scores, functional scores, and MRI data will be obtained pre-operatively and compared to the same data collected 1 year post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Burks, MD, Principal Investigator — University of Utah Orthopedics Center
Locations (1):
- University of Utah Orthopedics Center, Salt Lake City, Utah, United States